CLINICAL TRIAL: NCT03971591
Title: Men Moving Forward: A Lifestyle Program for African-American Prostate Cancer Survivors
Acronym: MMF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Loyola University Chicago (Other); Marquette University (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Melinda Stolley, Associate Director for Cancer Prevention and Control, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00031416
Record Dates: First submitted 2019-05-09; First posted 2019-06-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a guided or self-guided lifestyle intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Lifestyle program (Experimental): The Intervention will be conducted in cohorts of 15-20. We anticipate there will be 5-6 cohorts over the course of the study. Men assigned to the Guided Lifestyle Program will participate in twice weekly sessions - the first weekly session will be 120 minutes in length with the first hour addressing lifestyle change education and strategies, the second hour will be supervised exercise with strength training. The second weekly session will be a one-hour supervised exercise session with strength training. Men will also receive 2-3 text messages weekly. They will also receive a participant informational binder with health and exercise information and tools as directed by ACS nutrition and physical activity guidelines.
  Interventions: Behavioral: Immediate Guided Lifestyle Program Intervention
- Waitlist Control (Other): In the waitlist control arm, the men will not receive any intervention for 16-weeks. After the 16-week assessment, men randomized to this arm will crossover to the intervention arm.
  Interventions: Behavioral: Immediate Guided Lifestyle Program Intervention

INTERVENTIONS:
Behavioral: Immediate Guided Lifestyle Program Intervention — The Guided Lifestyle Program will receive sessions that meet twice weekly and 2-3 text messages weekly. They will also receive a participant informational binder with health and exercise information and tools as directed by ACS nutrition and physical activity guidelines.

SUMMARY:
This study will examine the efficacy of Men Moving Forward (MMF), a four-month community-based lifestyle intervention designed for AA PC survivors. MMF is rooted in the evidence-based Moving Forward lifestyle intervention developed with and for AA breast cancer survivors. This intervention was adapted in collaboration with AA PC survivors. It will offer twice weekly sessions aimed at supporting adherence to the ACS nutrition and physical activity guidelines to promote improved body composition (i.e., decreased adiposity, increased lean mass).

DETAILED DESCRIPTION:
Aim 1. To examine the efficacy of the Men Moving Forward guided intervention, as compared to a self-guided control intervention, in producing significant post-intervention changes in body composition in 200 AA PC survivors.

Hypothesis: Men randomized to the guided arm will exhibit significant post-intervention decreases in adiposity and increases in lean body mass compared to men randomized to the control arm.

Aim 2. To investigate the effects of participation in the Men Moving Forward guided intervention on health behaviors and quality of life outcomes.

Hypothesis: Men in the guided program will exhibit increased intake of fruits and vegetables and decreased intake of red meat/processed meat, greater levels of physical activity (minutes per week and #times/wk resistance training) and improved quality of life (targeting physical function, social isolation, sexual functioning) compared to men in the control arm.

Aim 3. To explore the effects of the intervention program on blood pressure, blood lipids, fasting glucose, and biomarkers associated with comorbidities and carcinogenesis (i.e adiponectin, leptin, C-peptide, IGF-1, IGFBP-3, C-Reactive Protein, estradiol, testosterone and sex hormone binding globulin)

Hypothesis: Men in the guided arm will exhibit greater improvements in biomarkers associated with chronic disease and carcionogenesis compared to men in the self-guided control arm.

Men Moving Forward supports PC survivors in adopting physical activity and eating patterns that will improve their body composition, bolster QOL and reduce risk for comorbidities and, potentially, PC recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Self-identify as Black or African American
* Diagnosed with non-metastatic Prostate Cancer (cancer that has NOT spread elsewhere in the body)
* Completed all treatments (including Androgen Deprivation Therapy) at least six months prior to enrollment
* BMI > 25 kg/m2
* Able to participate in moderate physical activity as assessed by healthcare provider
* Exercise less than the ACS recommended guideline of 150 min/week or 30 min/day.
* Fruit and vegetable consumption is less than 5 servings each day.
* Lift Weights or engage in strength training less than twice a week.
* Can walk continuously for 5 minutes without stopping because of pain or shortness of breath.
* Have access to a mobile phone
* Approval from Primary Care Provider/Medical Oncologist
* Available to attend intervention

Exclusion Criteria:

* • Does not meet the Inclusion Criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male Prostate Cancer study participants
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in body composition | Change from Baseline to 4 month
  Ratio of percent lean mass to percent adiposity as measured by DEXA. More lean mass and less adiposity is favorable.
Change in body composition | Change from Baseline to 12 month
  Ratio of percent lean mass to percent adiposity as measured by DEXA. More lean mass and less adiposity is favorable.
Increase in intake of fruits and vegetables | Change from Baseline to 4 month
  VioScreen's dietary analysis of self reported food consumption
Increase in intake of fruits and vegetables | Change from Baseline to 12 month
  VioScreen's dietary analysis of self reported food consumption
Decrease of intake of red meat/processed meat | Change from Baseline to 4 month
  VioScreen's dietary analysis of self reported food consumption
Decrease of intake of red meat/processed meat | Change from Baseline to 12 month
  VioScreen's dietary analysis of self reported food consumption
Increase in levels of physical activity- minutes per week | Change from Baseline to 4 month
  Change of ActiGraph monitored activity
Increase in levels of physical activity- minutes per week | Change from Baseline to 12 month
  Change of ActiGraph monitored activity
Increase in levels of physical activity- #times per week | Change from Baseline to 4 month
  Change of ActiGraph monitored activity
Increase in levels of physical activity- #times per week | Change from Baseline to 12 month
  Change of ActiGraph monitored activity
Increase in resistance training- Lower extremity strength | Change from Baseline to 4 month
  Isokinetic dynamometer (HUMAC Norm, Stoughton, MA).
Increase in resistance training- Lower extremity strength | Change from Baseline to 12 month
  Isokinetic dynamometer (HUMAC Norm, Stoughton, MA).
Increase in resistance training- Handgrip strength | Change from Baseline to 4 month
  Takei 5401 Hand Grip Digital Dynamometer
Increase in resistance training- Handgrip strength | Change from Baseline to 12 month
  Takei 5401 Hand Grip Digital Dynamometer
Increase in resistance training- Strength and endurance | Change from Baseline to 4 month
  30-Second Chair Stand (Sit to Stand)
Increase in resistance training- Strength and endurance | Change from Baseline to 12 month
  30-Second Chair Stand (Sit to Stand)
Change in Quality of Life- PROMIS | Change from Baseline to 4 month
  PROMIS T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. PROMIS measures physical function, depression, anxiety, fatigue, sleep disturbance, social roles, pain interference, social isolation, cognitive function, support, self-efficacy and sexual function.
Change in Quality of Life-PROMIS | Change from Baseline to 4 month
  PROMIS T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. PROMIS measures physical function, depression, anxiety, fatigue, sleep disturbance, social roles, pain interference, social isolation, cognitive function, support, self-efficacy and sexual function.
Change in Urban life stress inventory- Crisys | Change from Baseline to 4 month
  Measure change of mean in positive/negative/neutral and resolved/ongoing
Change in Urban life stress inventory-Crisys | Change from Baseline to 12 month
  Measure change of mean in positive/negative/neutral and resolved/ongoing
Changes in Blood Pressure | Change from Baseline to 4 month
  Participants blood pressure will be measured using a digital, automated unit
Change in Blood Pressure | Change from Baseline to 12 month
  Participants blood pressure will be measured using a digital, automated unit
Change in Biomarkers- Hemoglobin | Change from Baseline to 4 month
  Hemoglobin blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Hemoglobin | Change from Baseline to 12 month
  Hemoglobin blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- A1C | Change from Baseline to 4 month
  A1C blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- A1C | Change from Baseline to 12 month
  A1C blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- Hormones-Testosterone | Change from Baseline to 4 month
  Testosterone blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- Hormones-Testosterone | Change from Baseline to 12 month
  Testosterone blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- Hormones- Estradiol | Change from Baseline to 4 month
  Estradiol blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- Hormones- Estradiol | Change from Baseline to 12 month
  Estradiol blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- Hormones- SHBG | Change from Baseline to 4 month
  SHBG blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- Hormones- SHBG | Change from Baseline to 12 month
  SHBG blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Adipokines- Leptin | Change from Baseline to 4 month
  Leptin blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Adipokines- Leptin | Change from Baseline to 12 month
  Leptin,blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Adipokines-Adiponectin | Change from Baseline to 4 month
  Adiponectin blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Adipokines-Adiponectin | Change from Baseline to 12 month
  Adiponectin blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Inflammation- IL-6 | Change from Baseline to 4 month
  IL-6 blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Inflammation- IL-6 | Change from Baseline to 12 month
  IL-6 blood test measured by Wisconsin Diagnostic Laboratory Wisconsin
Change in Biomarkers-Inflammation-TNFα | Change from Baseline to 4 month
  TNFα blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Inflammation-TNFα | Change from Baseline to 12 month
  TNFα blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Insulin Resistance-C-Peptide | Change from Baseline to 4 month
  C-Peptide blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Insulin Resistance- C-Peptide | Change from Baseline to 12 month
  C-Peptide blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Insulin Resistance-IGF-1 | Change from Baseline to 4 month
  IGF-1 blood test measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers Insulin Resistance-IGF-1 | Change from Baseline to 12 month
  IGF-1 blood test measured by Wisconsin Diagnostic Laboratory

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Awoyinka I, Sheean P, Papanek P, Flynn KE, Bylow K, Kilari D, Gann P, Banerjee A, Stolley M. Study design and methodologies for the men moving forward lifestyle intervention trial with black prostate cancer survivors. Contemp Clin Trials. 2025 Dec 24;161:108205. doi: 10.1016/j.cct.2025.108205. Online ahead of print. PMID 41453520